CLINICAL TRIAL: NCT01109758
Title: Effects of Fenofibrate on Gene Expression Activity and DNA Methylation Profile in Circulating Monocytes of Healthy Volunteers
Brief Title: Effects of Fenofibrate on Gene Expression in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Claire Nee, Solvay Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S282.1.002; 2007-006147-52 (EudraCT Number)
Record Dates: First submitted 2010-04-12; First posted 2010-04-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Fenofibrate; Gene Expression; DNA methylation
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — 145 mg

SUMMARY:
The purpose of this study is to assess how fenofibrate modify gene expression in circulating monocytes of healthy volunteers after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* To be aged 40-65 years,
* To be post menopausal female not receiving hormone replacement therapy,
* To have normal homocysteine, folate and vitamin B12 levels at baseline (results available for initiation of treatment),
* To be in good health as determined by medical history, physical examination, ECG, vital signs, serum/urine biochemistry and hematology.

Exclusion Criteria:

* Subjects with clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, neurologic/psychiatric or emotional, respiratory, urogenital, hematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatologic/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, (drug) allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking the study medication,
* Subjects who have been treated with fenofibrate in a previous study,
* Subjects who have taken a single dose of an investigational drug within 30 days or multiple doses of any investigational drug within 60 days prior to dosing

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change of gene activity of markers in circulating monocytes between Baseline and 6 weeks of fenofibrate treatment | Between Baseline and 6 weeks
  The calculation is the difference between the gene expression intensity after 6 weeks of treatment and the gene expression intensity at Baseline
DNA methylation pattern | 6 weeks

SECONDARY OUTCOMES:
Fenofibric acid levels | 6 weeks
urinary protein profile | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, London, United Kingdom